CLINICAL TRIAL: NCT01478100
Title: Virtual Coronary Intervention and Non-invasive Fractional Flow Reserve (FFR)
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Bon-Kwon Koo, Associate Professor of Medicine, Seoul National University Hospital
Other Study IDs: H-1109-106-379
Record Dates: First submitted 2011-11-20; First posted 2011-11-23 (Estimated); Last update posted 2011-11-23 (Estimated); Status verified 2011-11

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease; CT; Computational flow dynamics
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators examined the feasibility of treatment planning using virtual coronary revascularization and fractional flow reserve (FFR) CT before the invasive procedures.

ELIGIBILITY:
Inclusion Criteria:

* Significant stenosis at CT angiography
* Normal ejection fraction on echocardiography
* Informed consented patient

Exclusion Criteria:

* Total occlusion and collateral flow to target vessel
* AV conduction abnormality
* Left ventricular hypertrophy
* Significant valvular heart or primary myocardial disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: From the DISCOVER-FLOW study 20 patients with available post-intervention FFR were included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2011-10; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Kim KH, Doh JH, Koo BK, Min JK, Erglis A, Yang HM, Park KW, Lee HY, Kang HJ, Kim YJ, Lee SY, Kim HS. A novel noninvasive technology for treatment planning using virtual coronary stenting and computed tomography-derived computed fractional flow reserve. JACC Cardiovasc Interv. 2014 Jan;7(1):72-8. doi: 10.1016/j.jcin.2013.05.024. Epub 2013 Dec 11. PMID 24332418